CLINICAL TRIAL: NCT03845400
Title: An Observational, Non-interventional, Study of Patients With Hereditary Angioedema in the United States and Canada (EMPOWER Study)
Brief Title: A Study of Lanadelumab in Persons With Hereditary Angioedema (HAE) Type I or II in North America
Acronym: EMPOWER
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP643-403; TAK-743-403 (Other: Takeda Development Center Americas)
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type I or Type II HAE Participants: Participants with Type I or Type II HAE will be followed for 24 or 36 months depending upon enrollment date. Data collection will cease at the end of follow-up period, at the time of withdrawal, lost to follow-up, or death whichever comes first.

SUMMARY:
The main aim of this study is to compare the HAE attack rate before and after lanadelumab treatment was started in persons with Hereditary Angioedeme Type I or II.

Data from participants will be collected for at least 24 months. Participants will report information in a smartphone application at study start and then every 3 months until the study ends; data will also be collected by the study doctor during routine clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written, signed, and dated (personally or via a legally-authorized representative) informed consent/and assent as applicable to participate in the study. Expression of understanding and agreement by fully informed parent(s) or legal guardian is required to permit the investigator to enroll a child in this study. The choice of the terms parental consent or parental permission in different regions may reflect local legal/regulatory and ethical considerations.
* Diagnosis of HAE Type I or Type II.
* Ability to use a mobile device for data collection in the study.

Exclusion Criteria:

* Participation in any interventional clinical trial at the time of enrollment.
* Unable to provide written, signed, and dated informed consent/assent.
* Investigator believes that the participant is not a suitable candidate for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a diagnosis of Type I or Type II HAE.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Number of Hereditary Angioedema (HAE) Attacks | From enrollment up to 36 months
  Number of HAE attacks before and after lanadelumab initiation will be reported.

SECONDARY OUTCOMES:
Dose of Lanadelumab Injections | From enrollment up to 36 months
  Dose of lanadelumab injections used during the study will be reported.
Frequency of Lanadelumab Injections | From enrollment up to 36 months
  Frequency of lanadelumab injections during the study will be reported.
Proportion of Injections Based on the Type of Administration of Lanadelumab | From enrollment up to 36 months
  Proportion of injections based on the type of administration of lanadelumab (self, caregiver, health care provider [HCP], other) will be reported.
Time From Diagnosis to Lanadelumab Initiation | From enrollment up to 36 months
  Time from diagnosis of HAE attack(s) to lanadelumab treatment initiation will be reported.
Proportion of Participants who Discontinue Lanadelumab | From enrollment up to 36 months
  Discontinuation is defined as no documented lanadelumab use after at least 2 missing consecutive doses after the last date of injection, or documented as treatment discontinued by the physician. Proportion of participants who discontinue lanadelumab treatment will be reported.
Number of Lanadelumab Injections Before Discontinuation per Reason for Injection | From enrollment up to 36 months
  Discontinuation is defined as no documented lanadelumab use after at least 2 missing consecutive doses after the last date of injection, or documented as treatment discontinued by the physician. Number of injections administered by participant before discontinuation per reason for injection will be reported.
Number of Hospitalizations due to Hereditary Angioedema (HAE) Attack(s) | From enrollment up to 36 months
  Number of hospitalizations due to HAE attack(s) will be reported.
Number of Emergency Room (ER) Visits due to Hereditary Angioedema (HAE) Attack(s) | From enrollment up to 36 months
  Number of emergency room (ER) visits due to HAE attack(s) will be reported.
Number of Physician Visits due to Hereditary Angioedema (HAE) Attack(s) | From enrollment up to 36 months
  Number of physician visits due to HAE attack(s) will be reported.
Rescue Medications Taken at Time of Hereditary Angioedema (HAE) Attack(s) | From enrollment up to 36 months
  Number, type of rescue medications taken by the participants at the time of HAE attack(s) per the type of administration (self, caregiver, HCP, other) will be reported.
Hereditary Angioedema (HAE) Attack Control Score Before and After Lanadelumab Initiation, as Measured by the Angioedema Control Test (AECT) | From enrollment up to 36 months (every 3 months)
  AECT is a questionnaire and not a validated patient-reported outcome (PRO). HAE control score is evaluated as frequency of answers [very often, often, sometimes, seldom, not at all] to the following questions at record closest to enrollment date): 1. In the last 3 months, how often have you had angioedema? 2. In the last 3 months, how much has your quality of life been affected by angioedema? 3. In the last 3 months, how much has the unpredictability of your angioedema bothered you? 4. In the last 3 months, how well has your angioedema been controlled by your therapy?
Angioedema Quality of Life (AE-QoL) Score | From enrollment up to 36 months (every 3 months)
  The AE-QoL is developed to measure health-related quality of life (HRQoL) impairment in participants with recurrent angioedema. It is a self-administered PRO designed for adults aged 18 years and older with a recall period of 4 weeks. There are 17 items across 4 domains: functioning (4 items), fatigue/mood (5 items), fears/shame (6 items), and food (2 items). Responses use a 5-point Likert scale ranging from 'never' to 'very often.' Global scores range from 0 to 100 and scores by domains range from 0 to 100.
Work Productivity and Activity Impairment: General Health (WPAI:GH) Score | From enrollment up to 36 months (every 3 months)
  The WPAI:GH is a generic questionnaire to measure the effect of general health and symptom severity on work productivity and regular activities during the past 7 days. It can be self- or interviewer-administered to adults aged 18 years or older. This 6-item PRO covers work (5 items) and daily activities (1 item) using yes/no or numerical answers (number of hours). WPAI:GH outcomes are expressed as impairment percentages. An overall work productivity score (health or symptom) [%0WP], is calculated by multiplying the percentage of work time spent working (health or symptom) [% WTW] by the percentage productivity at work (health or symptom) [%PW]: %0WP = %WTW * %PW.
Treatment Satisfaction (TSQM-9) Score | From enrollment up to 36 months (every 3 months)
  The TSQM is a generic questionnaire to measure participants' satisfaction with medication using yes/no and 5- or 7- point Likert scale response options. It is a self-administered PRO designed for adults aged 18 years or older with a recall period of 2 to 3 weeks, or since the last medication use. Version TSQM-9 includes 3 domains: effectiveness (3 items), convenience (3 items), and global satisfaction scale (3 items). Scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (29):
- United States (23):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of South Florida Asthma, Allergy & Immunology, Tampa, Florida
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Institute for Asthma & Allergy - Chevy Chase, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mid West Immunology Clinic, Plymouth, Minnesota
  - Washington University, St Louis, Missouri
  - Riverside Medical Group, Belleville, Belleville, New Jersey
  - Jay M Kashkin, MD Allergy, Asthma and Immunology, Fair Lawn, New Jersey
  - Mount Sinai, New York, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Duke Asthma, Allergy & Airway Center, Durham, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Portland Clinical Research/AAIM Care, Happy Valley, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington
- Canada (5):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - McMaster University Health Sciences Center, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CHUM Hôtel-Dieu, Montreal, Quebec
  - Clinique Specialisée en Allergie de la Capitale, Québec
- Rafael H Zaragoza-Urdaz, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Betschel SD, Chapdelaine H, Gagnon R, Goodyear MD, Keith PK, El-Zoeiby A, Khutoryansky N, Castaner DN. Long-term effectiveness and safety of lanadelumab in Canadian patients with hereditary angioedema: a subanalysis of the EMPOWER study. Allergy Asthma Clin Immunol. 2026 Jan 21. doi: 10.1186/s13223-025-01007-9. Online ahead of print. PMID 41566486
- [Derived] Zanichelli A, Wuillemin WA, Aygoren-Pursun E, Banerji A, Busse PJ, Betschel SD, Cancian M, Gagnon R, Goodyear MD, Kinaciyan T, Kessel A, Magerl M, Recke A, Wedner HJ, Estepan DN, Watt M, Andresen I, Juethner S, Khutoryansky N, Martinez-Saguer I. Lanadelumab's impact on hereditary angioedema control and quality of life across disease activity subgroups: Real-world evidence. Ann Allergy Asthma Immunol. 2025 Nov;135(5):560-569.e2. doi: 10.1016/j.anai.2025.07.025. Epub 2025 Sep 6. PMID 40769455
- [Derived] Bernstein JA, Betschel SD, Busse PJ, Banerji A, Wedner HJ, Manning M, Zaragoza-Urdaz RH, Anderson J, Gagnon R, Baptist AP, Soteres D, Lumry WR, Craig T, Petroni D, Hsu FI, Nova Estepan D, Juethner S, Watt M, Khutoryansky N, Zuraw BL; EMPOWER Investigators. Sustained Effectiveness, Tolerability, and Safety of Long-Term Prophylaxis with Lanadelumab in Hereditary Angioedema: The Prospective, Phase 4, Noninterventional EMPOWER Real-World Study. Adv Ther. 2025 Aug;42(8):3882-3901. doi: 10.1007/s12325-025-03226-3. Epub 2025 Jun 12. PMID 40504359
- [Derived] Tachdjian R, Banerji A, Busse PJ, Agmon-Levin N, Anderson J, Cancian M, Spadaro G, Enciu C, Estepan DN, Khutoryansky N, Jain S, Recke A. Effective long-term prophylaxis with lanadelumab in adolescents with hereditary angioedema: EMPOWER/ENABLE. Pediatr Allergy Immunol. 2025 Apr;36(4):e70072. doi: 10.1111/pai.70072. PMID 40171989
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab47320